CLINICAL TRIAL: NCT04084925
Title: Is HOMA-IR(Homeostatic Model Assessment for Insulin Resistance) a Potential Screening Test for Non-alcoholic Fatty Liver Disease in Adults With Type 2 DM?
Brief Title: HOMA-IR as a Screening Test in NAFLD
Status: Completed | Type: Observational
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Ahmed Abdelkawi Hammad, Lecturer of internal medicine-Faculty of medicine -Fayoum university, Fayoum University
Other Study IDs: M258
Record Dates: First submitted 2019-09-03; First posted 2019-09-10 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: NAFLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diabetics with NAFLD: Diabetics whose abdominal ultrasound showed that they have NAFLD
- Diabetics without NAFLD: Diabetics whose abdominal ultrasound showed that they do not have NAFLD

SUMMARY:
The aim of this study is to evaluate the role of HOMA-IR in diagnosis of NAFLD in patients with type 2 DM.

DETAILED DESCRIPTION:
this study is a retrospective cohort study included 100 patients with type 2 DM from the outpatient clinic of internal medicine department at Fayoum University Hospital. They were divided into two equal groups according to the presence of NAFLD by ultrasound. All patients were subjected to history taking, clinical examination and investigations which included: ALT, AST, total cholesterol, TG, FBG and fasting insulin level,HOMA-IR(Homeostatic Model Assessment for Insulin Resistance) assessment.

ELIGIBILITY:
Inclusion Criteria:

- Diabetes obesity

Exclusion Criteria:

* use of alcohol

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with type 2 diabetes mellitus from the outpatient clinic of internal medicine department at Fayoum University Hospital
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-06-20 (Actual); Study Completion 2018-12-20 (Actual)

PRIMARY OUTCOMES:
The correlation between HOMA-IF and NAFLD | 6 months
  Find a statistically significant correlation between HOMA IR and NAFLD in diabetics

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed A Mashaheet, MD, Study Director — Faculty of medicine Fayoum university
Locations (1):
- Fayoum university hospital, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: Undecided